CLINICAL TRIAL: NCT01699724
Title: Phase 1, Open-Label, Randomized, Single-Dose, 3-Way Crossover Assessing Bioequivalence Of Zoloft ODT 50 Mg Under Fasting Condition With And Without Water To Jzoloft Tablet 50 Mg Under Fasting Condition With Water In Healthy Japanese Subjects
Brief Title: Bioequivalence Of Zoloft ODT To Jzoloft In Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A0501098
Record Dates: First submitted 2012-09-18; First posted 2012-10-04 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: JZoloft; Sertraline hydrochloride; ODT; bioequivalence
MeSH Terms: interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- JZoloft (Active Comparator): Oral tablet of sertraline hydrochloride (Japanese commercial tablet: JZoloft ® tablet) 50 mg as a single oral dose under fasted conditions
  Interventions: Drug: JZoloft
- ODT without water (Experimental): sertraline ODT 50 mg without water as a single oral dose under fasted conditions
  Interventions: Drug: sertraline ODT
- ODT with water (Experimental): sertraline ODT 50 mg with water as a single oral dose under fasted conditions
  Interventions: Drug: sertraline ODT

INTERVENTIONS:
Drug: JZoloft — 50 mg tablet on Day 1 of each period
  Other Names: sertraline hydrochloride
  Arms: JZoloft
Drug: sertraline ODT — 50 mg tablet on Day 1 of each period
  Arms: ODT without water
Drug: sertraline ODT — 50 mg tablet on Day 1 of each period
  Arms: ODT with water

SUMMARY:
The purpose of this study is to assess the bioequivalence of Zoloft ODT 50 mg with and without water to Japanese commercial oral tablet of JZoloft 50 mg under fasting condition with water in Healthy Japanese Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese subjects between the ages of 20 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Significant psychiatric disorder, recurrent episodes of severe depression, or subjects with serious suicidal risk per criteria.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of nonhormonal contraception as outlined in this protocol from at least 14 days prior to the first dose of study medication and for 28 days after the last dose of study medication.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
AUC from zero to the last sampling point (AUCt) of sertraline after dose of sertraline ODT 50 mg without water to Japanese commercial oral tablet of JZoloft 50 mg under fasted conditions | 0, 1, 2, 4, 6, 7, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
Maximum plasma concentration (Cmax) of sertraline after dose of sertraline ODT 50 mg without water to Japanese commercial oral tablet of JZoloft 50 mg under fasted conditions | 0, 1, 2, 4, 6, 7, 8, 10, 12, 24, 36, 48 and 72 hours post-dose

SECONDARY OUTCOMES:
Cmax and AUCt of sertraline after dose of sertraline ODT 50 mg with water to Japanese commercial oral tablet of JZoloft 50 mg under fasted conditions | 0, 1, 2, 4, 6, 7, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
Time of maximum plasma concentration of sertraline ODT 50 mg with water to Japanese commercial oral tablet of JZoloft 50 mg under fasted conditions | 0, 1, 2, 4, 6, 7, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
AUC from zero to infinity or last measurable concentration of sertraline after dose of sertraline ODT 50 mg with and without water to Japanese commercial oral tablet of JZoloft 50 mg under fasted conditions | 0, 1, 2, 4, 6, 7, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
Terminal elimination rate constant (kel), half-life (t½) and mean residence time (MRT) of sertraline ODT 50 mg with and without water to Japanese commercial oral tablet of JZoloft 50 mg under fasted conditions | 0, 1, 2, 4, 6, 7, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
Safety laboratory tests, vital signs, and adverse events (AEs) | From Periods 1 to 3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Hachioji-shi, Tokyo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0501098&StudyName=Bioequivalence%20Of%20Zoloft%20ODT%20To%20Jzoloft%20In%20Healthy%20Japanese%20Subjects